CLINICAL TRIAL: NCT06174311
Title: The Effectiveness of Cognitive Bias Modification on Intolerance of Uncertainty: A Randomized Controlled Trial
Brief Title: The Effectiveness of Cognitive Bias Modification on Intolerance of Uncertainty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Selin Dumlu Gündoğan, Clinical Psychology Graduate Student, Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SGundogan; CGokdag (Other: ManisaCelalBayarU); YMeralOgutcu (Other: IzmirUEcon); EYuvruk (Other: MuglaSKU)
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Intolerance to Uncertainty
Keywords: Intolerance to Uncertainty; Cognitive Bias Modification

STUDY DESIGN:
Intervention Model Description: Condition 1: Cognitive Bias Modification for active group
  Condition 2: Cognitive Bias Modification for waitlist control group
Who Masked: Participant, Care Provider
Masking Description: Participants will be blinded to which condition they are assigned to. Participants will be assigned codes so that the care provider is also blinded to which condition the participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cognitive Bias Modification (Experimental): Based on the outcomes of pre-intervention measurements, 50 participants who score high on intolerance to uncertainty measurement will be chosen randomly to be included in this condition. This group of participants will receive three interventions targeting interpretation biases related to uncertainty, with each intervention administered at three-day intervals. Each session is scheduled to have an estimated duration of around 30 minutes.
  Interventions: Behavioral: Active Cognitive Bias Modification
- Control (Waitlist) Cognitive Bias Modification (No Intervention): The waitlist control group will not receive any interventions during the process. They will only undergo pre-test, post-test, and follow-up measurements. If they still wish to receive the intervention, it will be provided to them after the follow-up assessment.

INTERVENTIONS:
Behavioral: Active Cognitive Bias Modification — The intervention comprises three sessions and is provided online. Each session consists of two different tasks. To prevent order effects, these tasks will be presented to each participant in a random sequence. One of the tasks involves uncertain scenarios based on a scenario paradigm. At the end of these scenarios, participants will be asked to complete a missing letter in a word that in the scenario, followed by a comprehension question related to the scenario interpretation. Following each question, feedback will be provided regarding the correctness of the response. The other task is a word-sentence pair paradigm, where participants will be asked to assess whether these pairs are related, and feedback will also be provided.
  Arms: Active Cognitive Bias Modification

SUMMARY:
The current study aims to reduce the intolerance of uncertainty levels with an internet-based cognitive bias modification intervention in young adults with high levels of intolerance to uncertainty aged between 18 and 40. Furthermore, it aims to examine the intervention's effectiveness on their intolerance to uncertainty, positive and negative emotions, depression and anxiety symptoms, and repetitive thinking.

DETAILED DESCRIPTION:
Intolerance of uncertainty, a common factor in mental disorders (playing a transdiagnostic role), is critical to the development and maintenance of emotional problems (e.g., depression and anxiety) as it disrupts people's daily functioning. Studies have shown that intolerance of uncertainty is closely related to psychological problems, highlighting its importance for psychological interventions. Particularly considering the transdiagnostic nature of intolerance of uncertainty, attempting to reduce this trait in individuals also provides further intervention opportunities for various problems. Therefore, reducing intolerance of uncertainty is the focus of psychotherapy studies. The cognitive-behavioral conceptualization of intolerance of uncertainty emphasizes that people are unable to tolerate uncertainty because they misinterpret ambiguous situations in a biased manner, which leads to psychological problems. Accordingly, intervening in intolerance of uncertainty involves the modification of one's biased interpretations. At this point, Cognitive bias modification (CBM) is a method that involves paradigms in which a person is exposed to a series of stimuli to alter and reduce cognitive biases related to psychopathology. In recent years, the effectiveness of CBM in different psychological problems has been proven. In addition, current studies aim to reduce psychological symptoms through the use of CBM targeting transdiagnostic features and have shown promising results. Despite the importance of intolerance of uncertainty, only one study was found in the literature that examined the effect of CBM on intolerance to uncertainty in a randomized controlled design. In that study, it was concluded that a single-session CBM was successful in reducing intolerance to uncertainty by reducing interpretation biases in individuals. However, the study has some methodological shortcomings and requires further investigation in different samples. From this point of view, the present project aims to investigate the effectiveness of CBM on intolerance of uncertainty. The proposed project will examine the effect of internet-based CBM, focusing on interpretation bias related to uncertainty, on reducing intolerance of uncertainty and general psychological symptoms using self-report and behavioral measures in a randomized controlled design. In this way, the project aims to make a scientific contribution to the relatively limited literature in this area and to reduce participants' emotional symptoms by reducing their intolerance of uncertainty.

ELIGIBILITY:
Inclusion Criteria:

* Participants' willingness to participate in the CBM-I (Cognitive Bias Modification - Intervention)
* Having high levels of intolerance of uncertainty (receiving scores higher than the median of the initial sample by splitting the data based on the median)
* Having computer and internet access.

Exclusion Criteria:

* Being outside the targeted age range
* Having a psychiatric diagnosis and receiving current treatment
* Scoring psychotic questions and suicide questions above the midpoint on the Brief Symptom Scale
* Having color-blindness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Intolerance of Uncertainty Scale | Pre-intervention and up to 4 months
  The 12 items, rated on a 5-point scale (1= strongly disagree, 5= strongly agree), aim to measure individuals' intolerance of uncertainty levels. The scale provides two subscales (prospective and inhibitory) and a total score. High scores indicate a high level of intolerance of uncertainty.
Change in The Beads Task | Pre-intervention and up to 4 months
  This task is designed to behaviorally evaluate how and how quickly individuals make decisions in an uncertain situation (Huq et al., 1988; Phillips and Edwards, 1966).
Change in Interpretation Bias for Intolerance of Uncertainty | Pre-intervention and up to 4 months
  This task is used in Bias Modification for Interpretation studies to assess cognitive biases in participants before and after interventions. These tasks measure how individuals respond to stimuli similar to those they will encounter during the intervention phase, and the extent to which they make biased evaluations. The intervention in this project will consist of both a scenario task and a word-sentence association task. Therefore, in the interpretation bias task, participants' tendency to interpret uncertain scenarios and words negatively will be recorded. Participants will be presented with 10 scenarios, and they will be asked to assess the relatedness of four sentences for each scenario. Afterward, participants will be presented with 20 word-sentence pairs and expected to provide a yes or no response regarding whether they are related. The extent to which participants associate words signaling uncertainty with negative sentences will be used as a measure of interpretation bias.

SECONDARY OUTCOMES:
Change in Brief Symptom Measure | Pre-intervention and up to 4 months
  The scale consists of 25 items, rated on a 7-point scale (1= not at all, 7= extremely). The scale aims to assess individuals' general psychopathological symptoms. Obtaining a high score on the scale indicates a high level of symptomatology.
Change in Positive and Negative Affect Schedule | Pre-intervention and up to 4 months
  The scale consists of 20 emotion expressions, half of them positive and half negative, rated on a 5-point scale (1= very little or not at all, 5= very much). Participants are asked to assess how much they have felt these 20 emotions in the past week. The scale includes 10 emotion expressions related to Positive Emotions such as excited, alert, and 10 emotion expressions related to Negative Emotions such as distressed, guilty. Scores from these subscales indicate that a high level of positive emotion suggests contentment, while a high level of negative emotion indicates discontent.
Change in Repetitive Thinking Questionnaire | Pre-intervention and up to 4 months
  The scale comprises 10 items, rated on a 5-point scale (1= not at all true, 5= very true), and it is designed to measure individuals' general repetitive thinking tendencies as a trait. The scale provides a single score, with high scores indicating a high level of repetitive thinking tendencies.

OTHER OUTCOMES:
Feedback Form Questionnaire | Post-intervention (up to 4 months)
  The form includes questions for providing feedback about the intervention. In addition to the general evaluation items assessed with scales, it also incorporates open-ended questions allowing participants to provide feedback on aspects they like, dislike, and find boring, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir University of Economics, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is planned to add some files to the OSF (Open Science Framework) link created for the study.

REFERENCES:
- See also: OSF (Open Science Framework) file of the study — https://osf.io/xen9m/